CLINICAL TRIAL: NCT01506674
Title: Metabolomic in Critical Ill Patients
Status: Terminated | Type: Observational
Why Stopped: The study was terminated prematurely due to slow recruitment.
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, MD, Associate Professor, Università Vita-Salute San Raffaele
Other Study IDs: HSR CEmet
Record Dates: First submitted 2012-01-09; First posted 2012-01-10 (Estimated); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Metabolomic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- criticall ill patients

SUMMARY:
Analysis of blood, urinary, and intrathecal metabolites of critical ill patients will be checked for possible correlations between metabolomics patterns and patients' outcomes.

ELIGIBILITY:
Inclusion Criteria:

* patients with severe left or right ventricular dysfunction undergoing cardiac surgery
* patients undergoing ablation of ventricular tachycardia
* patients with febrile neutropenia after chemotherapy or allogeneic transplant for haematological diseases
* patients undergoing thoracoabdominal vascular surgery

Exclusion Criteria:

* pregnant women
* no written consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical ill patients
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Metabolomic patterns to identify poor outcome | hospital stay (approximately two weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Università Vita-Salute San Raffaele, Milan, Mi, Italy